CLINICAL TRIAL: NCT03531970
Title: Effect of Lidocaine/Dexamethasone on the Success of IANB in Patients With Irreversible Pulpitis
Brief Title: Effect of Lidocaine/Dexamethasone on the Success of IANB
Acronym: IANB
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Masoud Saatchi, DDS MSc, Professor of Endodontics, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 396731
Record Dates: First submitted 2018-05-02; First posted 2018-05-22 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Local Anesthesia
Keywords: inferior alveolar nerve block; irreversible pulpitis; local anesthesia; dexamethasone
MeSH Terms: interventions — Lidocaine; Epinephrine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Experimental): lidocaine & Dexamethasone
  Interventions: Drug: 2% lidocaine with 1:80,000 epinephrine; Drug: Dexamethasone
- Non-dexamethasone (Placebo Comparator): lidocaine & Placebo
  Interventions: Drug: 2% lidocaine with 1:80,000 epinephrine; Drug: Placebo

INTERVENTIONS:
Drug: 2% lidocaine with 1:80,000 epinephrine — Anesthetic solution
  Other Names: lidocaine (2% Persocaine-E; Daroupakhsh, Tehran, Iran)
Drug: Dexamethasone — Corticostroide
  Other Names: Dexamethasone (Caspian Tamin Pharmaceutical Co, Rasht, Iran)
  Arms: Dexamethasone
Drug: Placebo — Placebo
  Other Names: sterile distilled water (Samen Pharmaceutical Co, Iran)
  Arms: Non-dexamethasone

SUMMARY:
The purpose of this prospective, randomized, double-blind study was to compare the success rate of IAN block injection carried out with two cartridges of 2% lidocaine with 1:80000 epinephrine each combined with 0.2 ml dexamethasone versus two cartridges of 2% lidocaine with 1:80000 epinephrine each combined with 0.2 ml sterile distilled water for endodontic treatment of mandibular molars with symptomatic irreversible pulpitis.

DETAILED DESCRIPTION:
Several investigations have been carried out to demonstrate the effect of dexamethasone added to local anesthetics in regional block injections. These investigations shown that the addition of dexamethasone to local anaesthetics may prolong the duration of anesthesia and also results in a faster onset. It is hypothesized that dexamethasone added to lidocaine may affect the success rate of inferior alveolar nerve block

ELIGIBILITY:
Inclusion Criteria:

* vital mandibular molar tooth
* diagnosis of symptomatic irreversible pulpitis

Exclusion Criteria:

* younger than 18 years old
* history of significant medical conditions
* allergies to local anesthetics or sulfites
* pregnancy
* taking any medications that might influence anesthetic assessment
* active sites of pathosis in area of injection
* inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
success of IAN Block anesthesia for the Dexamethasone group | 15 minutes after the local anesthetic injection (at time of access cavity preparation)
  The success of the anesthesia was defined as the tooth without pain or with mild pain according to the Heft-Parker visual analog scale (HP-VAS ≤ 54). This scale is a 170-mm horizontal line, divided into 4 categories. No pain corresponded to 0 mm; mild pain was defined as >0 mm and 54 mm. Mild pain category included faint, weak and mild pain. A score >54 mm and <114 mm indicated moderate pain and included the descriptor of moderate pain. A score >54 mm and <114 mm indicated moderate pain and included the descriptor of moderate pain. Severe pain was defined as ≥114 mm. Severe pain was defined as strong, intense and maximum possible.
success of IAN Block anesthesia for the Non-dexamethasone group | 15 minutes after the local anesthetic injection (at time of access cavity preparation)
  The success of the anesthesia was defined as the tooth without pain or with mild pain according to the Heft-Parker visual analog scale (HP-VAS ≤ 54). This scale is a 170-mm horizontal line, divided into 4 categories. No pain corresponded to 0 mm; mild pain was defined as >0 mm and 54 mm. Mild pain category included faint, weak and mild pain. A score >54 mm and <114 mm indicated moderate pain and included the descriptor of moderate pain. A score >54 mm and <114 mm indicated moderate pain and included the descriptor of moderate pain. Severe pain was defined as ≥114 mm. Severe pain was defined as strong, intense and maximum possible.

SECONDARY OUTCOMES:
initial pain | Baseline
  rating the pain on Heft-Parker visual analog scale. This scale is a 170-mm horizontal line, divided into 4 categories. No pain corresponded to 0 mm; mild pain was defined as >0 mm and 54 mm. Mild pain category included faint, weak and mild pain. A score >54 mm and <114 mm indicated moderate pain and included the descriptor of moderate pain. A score >54 mm and <114 mm indicated moderate pain and included the descriptor of moderate pain. Severe pain was defined as ≥114 mm. Severe pain was defined as strong, intense and maximum possible.

CONTACTS AND LOCATIONS:
Overall Officials: Masoud Saatchi, Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Isfahan University of Medical Sciences, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: No